

| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Plan | Version Number: | 3.1 |
| | Effective Date: | 25-Nov-2021 |

# Statistical Analysis Plan

# **Study Title**

A prospective, multicenter, phase -IV study to assess the safety of fixed dose combination of dapagliflozin and saxagliptin in Indian Type 2 Diabetes Mellitus (T2D) patients

| Protocol/ Study Number : | D1683C00013 |
|--------------------------|-------------------------------------------------|
| Sponsor Name : | AstraZeneca Pharma India Limited |
| Sponsor Address : | AstraZeneca Pharma India Limited, |
| Y ~ | Block N1, 12th Floor, Manyata Embassy Business |
| | Park |
| | Rachenahalli, Outer Ring Road, Bangalore-560045 |
| Document Version : | 1.0 |
| Document Date : | 29-Jun-2022 |
| Author Name (s) : | PPD / |
| Author Name (3) | 0/. |
| Designation : | Biostatistician |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

# Table of Contents

| | Document Pag | e 2 of 71 |
|-----|-----------------------------------------------------|-----------|
| | 6.2 Study Hypothesis | 14 |
| | 6.1.2 Secondary Endpoint | 14 |
| | 6.1.1 Primary Endpoint | 14 |
| | 6.1 Study Endpoints | 14 |
| 6. | Study Analysis Strategy | 14 |
| | 5.5 Demographic Characteristics | |
| | 5.4 End Treatment | 13 |
| | 5.3 Disposition of Patients | |
| | 5.2 Decimal Point | |
| | 5.1 General Considerations | |
| | Patient Characteristics and Study Conduct Summaries | |
| | Sample Size and Power Calculations | |
| | 3.1 Safety population | |
| | Population Analysis Set | |
| | 2.5 Interim Analysis | |
| | 2.4 Blinding and Un-Blinding | |
| | 2.3 Randomization | |
| | 2.2.5 Study Plan | |
| | 2.2.4 Study Flow chart | |
| | 2.2.3 Exclusion Criteria | |
| | 2.2.2 Inclusion Criteria | |
| | 2.2.1 Study Design | |
| | 2.2 Study Description | |
| | 2.1.2 Secondary Objective | |
| | 2.1.1 Primary Objective | |
| | 2.1 Study Objective | |
| | Study Objective and Design | |
| | INTRODUCTION | |
| | ST OF ABBREVIATION | |
| | ST OF LISTING | |
| | ST OF TABLE | |
| 110 | ST OF TABLE | / |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

| ( | 5.3 Statstical Methods for Study Analsysis | . 14 |
|------------|--------------------------------------------|------|
| | 6.3.1 Primary Endpoint Analysis | |
| | 6.3.2 Secondary Endpoint Analysis | |
| <b>,</b> , | References | |
| 8. 1 | Mock Tables | .16 |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

# LIST OF TABLE

| Table 14.1.1.1. Patient Disposition in the Study (Enrolled Population) | 16 |
|---|---|
| Table 14.1.1.2. Summary of End Treatment (Safety Population) | 17 |
| Table 14.1.1.3. Summary of Analysis Population (Enrolled Population) | 18 |
| Table 14.1.2.1. Summary of Demographic Characteristics (Enrolled Population) | 19 |
| Table 14.1.2.2. Summary of Anthropometric Assessment (Safety Population) | 20 |
| Table 14.1.3. Summary of Medical and Surgical History (Safety Population) | 21 |
| Table 14.1.4. Summary of Urine Pregnancy Test (Safety Population) | 22 |
| Table 14.1.5. Summary of IP Medication Accountability (Safety Population) | 23 |
| Table 14.2.1. Analysis of change in HbA1c from baseline to Week 24 (Safety Population) | 24 |
| Table 14.2.2. Analysis of change in Weight from baseline to Week 24. (Safety Population) | 25 |
| Table 14.2.3. Analysis of change in Blood Pressure from baseline to Week 24. (Safety Population) | 26 |
| Table 14.2.4. Analysis of change in Fasting Plasma Glucose from baseline to Week 24. (Safety Population) | 27 |
| Table 14.2.5. Summary of HbA1c and Fasting Plasma Glucose (Safety Population) | 28 |
| Table 14.3.5. Summary of Hypoglycemic Event (Safety Population) | 29 |
| Table 14.3.1. Summary of Adverse Event (Safety Population) | 31 |
| Table 14.3.2. Summary of Adverse Event of special interest (Safety Population) | 33 |
| Table 14.3.3. Summary of Haematology Parameter (Safety Population) | 34 |
| Table 14.3.4. Summary of Clinical Chemistry Parameter (Safety Population) | 35 |
| Table 14.3.5. Summary of Urinalysis (Safety Population) | 36 |
| Table 14.3.6. Summary of Electrocardiogram (Safety Population) | 37 |
| Table 14.3.7. Summary of Vital Signs (Safety Population) | 38 |
| Table 14.3.8. Summary of Physical examination | 39 |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

# LIST OF LISTING

| Listing 16.2.1.1. Listing of Patients Informed Consent Details | 40 |
|---|---|
| Listing 16.2.1.2. Listing of Patients End of Treatment | 41 |
| Listing 16.2.1.3. Listing of Patients Study Completion | 42 |
| Listing 16.2.1.4. Listing of Analysis Population | 43 |
| Listing 16.2.2.1. Listing of Patients Demographics | 44 |
| Listing 16.2.2.2. Listing of Patients Anthropometric Assessment | 45 |
| Listing 16.2.3. Listing of Patients Medical History | 46 |
| Listing 16.2.4. Listing of Patients Urine Pregnancy test (Women of child bearing potential) | 47 |
| Listing 16.2.5.1. Listing of Patients IP Dispensing | 48 |
| Listing 16.2.5.2. Listing of Patients IP Medication Accountability | 49 |
| Listing 16.2.6.1. Listing of Patients HbA1c and Fasting Plasma Glucose | 50 |
| Listing 16.2.6.2. Listing of Patients Fasting Plasma Glucose | 51 |
| Listing 16.2.7.1. Listing of Patients Hypoglycaemic Event (Part I) | 52 |
| Listing 16.2.7.2. Listing of Patients Hypoglycaemic Event (Part II) | 53 |
| Listing 16.3.1.1. Listing of Patients Adverse Event Assessment | 54 |
| Listing 16.3.1.2. Listing of Patients Adverse Event | 55 |
| Listing 16.3.2. Listing of Patients Serious Adverse Event | 56 |
| Listing 16.3.3.1 Listing of Patients Haematology (WHOLE BLOOD) | 57 |
| Listing 16.3.3.2. Listing of Patients Clinical chemistry (Plasma / Serum) | 58 |
| Listing 16.3.3.3. Listing of Patients Urinalysis (Dipstick) | 59 |
| Listing 16.3.4. Listing of Patients Electrocardiogram (ECG) | 60 |
| Listing 16.3.5. Listing of Patients Vital Signs | 61 |
| Listing 16.3.6. Listing of Patients Physical Examination | 62 |
| Listing 16.3.7. Listing of Patients Other Assessment | 63 |
| Listing 16.3.8.1. Listing of Patients Urinary Tract Infection | 64 |
| Listing 16.3.8.2. Listing of Patients Genital Tract Infection | 65 |
| Listing 16.3.8.3. Listing of Patients Volume Depletion | 66 |
| Listing 16.3.8.4. Listing of Patients Diabetic Ketoacidosis | 67 |
| Listing 16.3.8.5. Listing of Patients Renal Events | 68 |
| Listing 16.3.8.6. Listing of Patients Hospitalization for Heart Failure | 69 |
| Listing 16.3.9.1. Listing of Patients Concomitant Medications | 70 |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

# LIST OF FIGURES

Not Applicable



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

# LIST OF ABBREVIATION

| Abbreviation | Term |
|---|---|
| AE | Adverse Event |
| ALP | Alkaline phosphatase |
| AST | Aspartate aminotransferase |
| BMI | Body Mass Index |
| CABG/PTCA | coronary artery bypass grafting/percutaneous transluminal coronary |
| | angioplasty |
| СК | Creatine kinase |
| CRF | Case Report Form (electronic/paper) |
| DAE | Discontinuation of Investigational Product due to Adverse Event |
| DKA | Diabetic ketoacidosis |
| EC | Ethics Committee, synonymous to Institutional Review Board (IRB) |
| | and Independent Ethics Committee (IEC) |
| ECG | Electrocardiogram |
| eGFR | Estimated Glomerular Filtration Rate |
| ESRD | End Stage Renal Disease |
| FBG | Fasting Blood Glucose |
| FDC | Fixed Dose Combination |
| FPG | Fasting Plasma Glucose |
| GCP | Good Clinical Practice |
| Hb | Hemoglobin |
| HbA1c | Glycated haemoglobin |
| ICH | International Council on Harmonisation |
| International Coordinating | If a study is conducted in several countries the International |
| investigator | Coordinating Investigator is the Investigator coordinating the |
| | investigators and/or activities internationally |
| IP | Investigational Product |
| IVRS | Interactive Voice Response System |
| IWRS | Interactive Web Response System |
| LIMS | Laboratory Information Management System |
| LSLV | Last Subject Last Visit |
| NYHA | New York Heart Association |
| OAE | Other Significant Adverse Event |
| PI | Principal Investigator |
| PPG | Post prandial Glucose |
| SAE | Serious Adverse Event |
| SBP | Systolic Blood Pressure |
| SGLT | Sodium Glucose Co transporter |
| SU | Sulphonylurea |
| T2DM | Type 2 Diabetes Mellitus |
| TIA | Transient Ischemic Attack |
| UPT | Urine Pregnancy Test |
| UTI | Urinary Tract Infection |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

#### 1. INTRODUCTION

The purpose of this document is to provide a description of the statistical methods and procedures to be implemented for the analysis of data from D1683C00013 study. This document is based on protocol V 3.0, 23 Sep 2020. The statistical planning and conduct of analysis of the data from this study will follow the principles defined in relevant International Council on Harmonisation (ICH)-E9 guidelines. Any change from the planned analysis as described in the protocol, are detailed here, and any differences described here supersede the analysis as presented in the protocol.

# 2. Study Objective and Design

# 2.1 Study Objective

#### 2.1.1 Primary Objective

To describe the adverse events profile of dapagliflozin + saxagliptin fixed dose combinations in Indian T2DM patients.

# 2.1.2 Secondary Objective

To describe the efficacy of dapagliflozin + saxagliptin fixed dose combination in Indian T2DM patient

#### 2.2 Study Description

## 2.2.1 Study Design

This is a prospective, multicenter, phase -IV study to assess the safety of fixed dose combination of dapagliflozin and saxagliptin in Indian Type 2 Diabetes Mellitus (T2D) patients.

Informed consent will be obtained from all the screened Patients prior to enrollment in the study. This study will include patients with T2DM.

This study is planned as prospective, multicentre, Phase-IV study on 200 patients in single arm open label study.



This is a 24-week open label prospective study. After eligibility check as per inclusion and exclusion criteria, patients will be recruited in the study and procedures as mentioned in below Section 2.2.5 will be performed at various scheduled visits.

#### 2.2.2 Inclusion Criteria

For inclusion in the study subjects should fulfil the following criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures according to local Indian procedure.

| Document | Proprietar | v and | Confid | lential | Document |
|---|---|---|---|---|---|
|---|---|---|---|---|---|



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

- 2. Male and female patients aged > 18 and above
- 3. Documented history of type 2 diabetes mellitus with HbA1c level >7.0% and ≤ 10% at screening visit
- Patients who are on a stable dose of antidiabetic drugs (including on Metformin dose between 1000-2000mg)
   in the past 3 months
- 5. Female subjects must be 1 year post-menopausal, surgically sterile, or using an acceptable method of contraception (an acceptable method of contraception is defined as a barrier method in conjunction with a spermicide) for the duration of the study (from the time they sign consent) to prevent pregnancy. In addition, oral contraceptives, approved contraceptive implant, long-term injectable contraception, intrauterine device, or tubal ligation are allowed. Oral contraception alone is not acceptable; additional barrier methods in conjunction with spermicide must be used.

#### 2.2.3 Exclusion Criteria

- 1. Known allergies or contraindication to the contents of the IP, dapagliflozin or saxagliptin tablets.
- 2. Active participation in another clinical study with IP and/or investigational device
- 3. For women only currently pregnant (confirmed with positive pregnancy test) or breastfeeding.
- 4. Type 1 diabetes mellitus.
- 5. Treatment with a SGLT2 inhibitor, GLP-1 agonist or DPP4 inhibitors at Visit 1 or 2
- 6. Patients with moderate to severe renal impairment (eGFR persistently <45 mL/min/1.73m<sup>2</sup> by CKD-EPI formula, or end-stage renal disease (ESRD) or 'Unstable or rapidly progressing renal disease
- 7. Patients with severe hepatic impairment (Child-Pugh class C)
- 8. History of pancreatitis or pancreatic surgery
- 9. Patients with a history of any malignancy
- 10. Patients with any of the following CV/Vascular Diseases within 3 months prior to signing the consent at enrolment, as assessed by the investigator:
  - Myocardial infarction.
  - Cardiac surgery or revascularization (CABG/PTCA).
  - Unstable angina.
  - Transient ischemic attack (TIA) or significant cerebrovascular disease.
  - Unstable or previously undiagnosed arrhythmia.
- 11. History of heart failure
- 12. Severe uncontrolled hypertension defined as systolic blood pressure ≥180 mm Hg and/or diastolic blood pressure ≥110 mm Hg at any visit up to randomisation



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

- 13. History of diabetic ketoacidosis
- 14. Any acute/chronic systemic infections
- 15. Recurrent urogenital infections
- 16. Patients at risk for volume depletion as judged by the investigator
- 17. Any condition which, in the judgment of the Investigator, may render the patient unable to complete the study or which may pose a significant risk to the patient or patient suspected or with confirmed poor protocol or medication compliance

# 2.2.4 Study Flow chart

Dapagliflozin 10|mg and Saxagliptin 5 mg Fixed Dose Combination



E = Enrollment, TC=Telephone Contact, EOT: End Of Treatment, EoS= End of Study

# 2.2.5 Study Plan

| | Visit 1 | Visit2 | Visit 3# | Visit 4# | Visit 5# | Visit 6# | Visit 7# | Visit 8# | Visit 9# | Visit10# |
|---|---|---|---|---|---|---|---|---|---|---|
| Assessments | Enrolment*<br>(-1 wk) | (0wk) | (1wk) | (4wk) | (8wk) | (12wk) | (16wk) | (20wk) | (24wk) | (26wk) |
| Window period<br>(Days) | (±5) | (±5) | (±2) | (±2) | (±5) | (±2) | (±5) | (±2) | (±5) | (±2) |
| Informed Consent | X | | | | | | | | | |
| Physical Exam | Х | Χ | | | X | | Х | | Х | Χ |
| Vital Signs | X | Χ | | | X | | X | | X | X |
| Eligibility Check | X | Х | | | | | | | | |
| HbA1c | Х | Х | | | Х | | Х | | Х | Χ |
| Fasting Plasma<br>Glucose<br>(FPG)*** | | Х | | | x | | х | | х | X |
| Weight & Height | | X | | | Х | | Х | | Х | X |
| Waist<br>Circumference | | Х | | | Х | | х | | Х | Х |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

| BMI (Body Mass<br>Index) | | х | | | x | | х | | х | х |
|--------------------------|---|---|---|---|---|---|---|---|---|---|
| Blood Pressure | | Х | | | X | | Х | | X | X |
| Safety labs | Х | Х | | | X | | Χ | | X | Χ |
| ECG | | X | | | | | X | | X | X |
| AE Assessment | | Х | X | Х | X | X | Х | Х | Х | X |
| Urinalysis | Х | Х | | | Х | | Х | | Х | Χ |
| UPT (WOCBP) | X | X | | | X | | X | | X | X |
| IP dispensation | | X | | | X | | | | | |
| IP accountability | | Х | Х | X | X | Х | X | | Х | X |

<sup>\*</sup>Enrolment and Visit 2 can coincide to enter patient into the study, #telephonic visit

#### 2.3 Randomization

Not Applicable

#### 2.4 Blinding and Un-Blinding

Not Applicable

#### 2.5 Interim Analysis

Not Applicable

# 3. Population Analysis Set

#### 3.1 Safety population

The safety analysis population will include all patients who sign the ICF and receive at least one dose of study medication.

The safety analysis population is also applicable to the efficacy analysis, and any efficacy measurements collected before the study medication discontinuation will be included. Last on treatment observation will be carried forward to impute the missing data at week 24.

# 4. Sample Size and Power Calculations

This is an India regulatory requirement study. Objective is to establish that FDC of Dapagliflozin 10mg / Saxagliptin 5 mg is a safe treatment option in Indian T2DM patients. This study is planned as prospective study on 200 patients in single arm open label study.

<sup>\*\*</sup> Subjects must be in a fasting state at least 8 hours prior to study visit.



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

# 5. Patient Characteristics and Study Conduct Summaries

#### 5.1 General Considerations

Statistical Analysis will be performed using SAS (version 9.4 or higher) software (SAS Institute Inc USA). Categorical variables will be summarized with the frequency and percentage of Patients in each category. Continuous variables will be summarized descriptively with the number of Patients, mean, standard deviation, minimum, median and maximum values.

#### 5.2 Decimal Point

Unless otherwise noted, means, median, will be presented to one decimal place more than the measured value, the same decimal as the measured value, percentages and confidence intervals will be presented to two decimal places and p-value will be presented to three decimal place. Percentages after zero counts will not be displayed and percentages equating to 100% will be presented as 100%, without any decimal places.

#### 5.3 Disposition of Patients

Patient disposition table will be based on all Enrolled Population who consented to participate in the study. The following summaries will be included in the disposition table: total number of Patients screened in the study, number of Patients who failed screening, number of Patient enrolled, number and percentage of Patients who completed the study and number and percentage of Patients who discontinued from the study with reason for discontinuation.

#### 5.4 End Treatment

Patient End Treatment table will be based on all Safety Population. The following summaries will be included in the End Treatment table: total number and percentage of Patient who Completed the Treatment and number and percentage of Patient who discontinued from the Treatment with Most appropriate reason for withdrawal/discontinuation of study

#### 5.5 Demographic Characteristics

Demographic and baseline characteristics will be summarized based on the Enrolled Population.

Descriptive summaries will be provided for the demographic and baseline characteristics. Demographic characteristics and baseline characteristics such as age, Gender and Race, etc. will be summarized and tabulated for Safety Population.

All the continuous variables will be summarized by n, mean, standard deviation, minimum, median and maximum values. All the categorical variables will be summarized as counts and percentages.



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

# 6. Study Analysis Strategy

# 6.1 Study Endpoints

# 6.1.1 Primary Endpoint

- Adverse Events (AEs) including Serious adverse events (SAEs), AEs leading to discontinuation (DAE) and
  adverse events of special interest (volume depletion, renal events, major hypoglycaemic events, fractures,
  urinary/genital tract infections, diabetic ketoacidosis, amputations and hospitalization for heart failure)
- Safety laboratory values
- Electrocardiogram (ECG)
- Vital Signs (pulse and BP)
- Physical examination

#### 6.1.2 Secondary Endpoint

- HbA1c change at week 24 compared to baseline
- Weight change at week 24 compared to baseline
- Systolic Blood Pressure (SBP) change at week 24 compared to baseline
- FPG change at week 24 compared to baseline

#### 6.2 Study Hypothesis

## Not Applicable

## 6.3 Statstical Methods for Study Analsysis

Statistical Analysis will be performed using SAS (version 9.4 or higher) software (SAS Institute Inc USA). Categorical variables will be summarized with the frequency and percentage of Patients in each category. Continuous variables will be summarized descriptively with the number of Patients, mean, standard deviation, minimum, median and maximum values.

#### 6.3.1 Primary Endpoint Analysis

The primary analysis for primary endpoint will be based on Safety Population.

Primary Endpoint evaluations will include adverse event monitoring, Safety Laboratory parameter, Electrocardiogram, VitalSigns and physical examinations.

Adverse Events (AEs) including Serious adverse events (SAEs), AEs leading to discontinuation (DAE) and adverse events of special interest (volume depletion, renal events, major hypoglycaemic events, fractures, urinary/genital tract



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

infections, diabetic ketoacidosis, amputations and hospitalization for heart failure) will be summarized using Frequency and percentages.

Safety laboratory Parameter data will be collected as per visit schedule. Observed values will be summarized descriptively (n, mean, median, standard deviation, minimum, and maximum values). A listing will be provided which contains data for each laboratory parameter.

Electrocardiogram parameters data will be collected as per visit schedule. Observed values will be summarized descriptively (n, mean, median, standard deviation, minimum, and maximum values). A listing will be provided which contains data for each Electrocardiogram parameter.

Vital Signs will be summarized based on the Safety population. Descriptive summaries will be provided for the Vital Signs. All the Categorical variables will be summarized with the frequency and percentage of Patients in each category. Continuous variables will be summarized descriptively with the number of Patients, mean, standard deviation, minimum, median and maximum values.

Physical Examination will be summarized based on the Safety populations. Descriptive summaries will be provided for the Physical Examination. All the categorical variables will be summarized as frequency and percentages.

#### 6.3.2 Secondary Endpoint Analysis

The Secondary analysis for Secodary endpoints will be based on Safety Population.

The safety analysis population is also applicable to the Secondary Endpoint analysis, and any Secondary Endpoint efficacy measurements collected before the study medication discontinuation will be included. Last on treatment observation will be carried forward to impute the missing data at week 24.

The Secondary endpoints (HbA1c, Weight, Blood Pressure and FPG) in this study is to evaluate the change from baseline to Post-baseline will be analysed using Paired t – test / Wilcoxon signed-rank test at 5% level of significance. Change from baseline will be determined as:

Change from Baseline = (Post-baseline - Baseline)

Percent Change Change from Baseline = ([Post-baseline - Baseline] / Baseline) X 100

## 7. References

- 1. ICH E3 Guideline\_International Council for Harmonisation
- 2. ICH E9; STATISTICAL PRINCIPLES FOR CLINICAL TRIALS



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

# 8. Mock Tables

Table 14.1.1.1. Patient Disposition in the Study (Enrolled Population)

| | N = xx |
|---------------------------------|------------|
| | n (%) |
| Patients Screened | xx |
| Screen Failures | xx |
| Patient Enrolled | xx |
| Patients Completed the study | xx (xx.xx) |
| Patients Discontinued the study | xx (xx.xx) |
| Reason for Discontinuation | |
| Withdrawal of Informed Consent | xx (xx.xx) |
| Discontinuation of the study | xx (xx.xx) |
| Other | xx (xx.xx) |
| Other 1 | xx (xx.xx) |
| Other 2 | xx (xx.xx) |

- The Capital "N" in the column header represents the total number of Enrolled Population.
- The small "n" in summary statistics represents the total number of Patients.
- Percentages in the "Patient completed the study" and "Patients Discontinued the study" rows are based on the total number of Enrolled Patients.
- Percentages in the "Reasons for Discontinuation" rows are based on the number of Patients Discontinued study.
- Note: Screened Patients are those who signed the informed consent
- Source :Listing 16.2.1.1 and Listing 16.2.1.3



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.1.1.2. Summary of End Treatment (Safety Population)

| | N = xx |
|---|---|
| | n (%) |
| Treatment with study drug discontinued prematurely | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| Reason for withdrawal/discontinuation of Study | |
| Voluntary discontinuation by the subject | xx (xx.xx) |
| Risk to subjects | xx (xx.xx) |
| Severe non-compliance to protocol | xx (xx.xx) |
| Incorrectly enrolled subjects | xx (xx.xx) |
| Adverse Event | xx (xx.xx) |
| Major and/or frequent hypoglycemic events | xx (xx.xx) |
| Diabetic Ketoacidosis | xx (xx.xx) |
| Acute renal insufficiency or worsened chronic renal insufficiency | xx (xx.xx) |
| Pregnancy | xx (xx.xx) |
| Lost to follow up | xx (xx.xx) |

- The Capital "N" in the column header represents the total number of Safety Population.
- The small "n" in summary statistics represents the total number of Patients.
- Percentages in the "Treatment with study drug discontinued prematurely" rows are based on the total number of Safety Patients.
- Percentages in the "Reasons for Withdrwal/Discontinuation of Treatment" rows are based on the number of Patients Treatment with study drug discontinued prematurely.
- Source :Listing 16.2.1.2



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.1.1.3. Summary of Analysis Population (Enrolled Population)

| | N = xx |
|-------------------|------------|
| | n (%) |
| Safety Population | xx (xx.xx) |

- The Capital "N" in the column header represents the total number of Enrolled Population.
- The small "n" in summary statistics represents the total number of Patients.
- Percentages in the "Safety Population" row is based on the total number of Enrolled Population.
- Safety Population: The Safety Population include all Patient who sign the ICF and receive at least one dose of study medication.



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.1.2.1. Summary of Demographic Characteristics (Enrolled Population)

| Demographic and Baseline Variables | N = xx |
|------------------------------------|----------------|
| Age (Years) | |
| n | Xx |
| Missing | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |
| Gender | |
| Male | xx (xx.xx) |
| Female | xx (xx.xx) |
| Missing | xx (xx.xx) |
| Race | |
| Asian | xx (xx.xx) |
| Other | xx (xx.xx) |
| Other 1 | xx (xx.xx) |
| Other n | xx (xx.xx) |

- The Capital "N" in the column header represents the total number of Enrolled Population.
- The small "n" in summary statistics represents the total number of Patients.
- Percentages are based on number of Enrolled Population.
- SD = Standard Deviation, min=minimum, max=maximum
- Source: Listing 16.2.2.1



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.1.2.2. Summary of Anthropometric Assessment (Safety Population)

| | N = xx |
|--------------------------|----------------|
| Visit x | |
| Height (cm) | |
| n | XX |
| Missing | XX |
| Mean (SD) | xx.x (xx.xx) |
| Median | XX.X |
| (min, max) | (xx.xx, xx.xx) |
| Weight (Kg) | |
| n | XX |
| Missing | XX |
| Mean (SD) | xx.x (xx.xx) |
| Median | XX.X |
| (min, max) | (xx.xx, xx.xx) |
| Waist circumference (cm) | |
| n | XX |
| Missing | XX |
| Mean (SD) | xx.x (xx.xx) |
| Median | XX.X |
| (min, max) | (xx.xx, xx.xx) |
| Body Mass Index (Kg/m²) | |
| n | XX |
| Missing | XX |
| Mean (SD) | xx.x (xx.xx) |
| Median | XX.X |
| (min, max) | (xx.xx, xx.xx) |

- The Capital "N" in the column header represents the total number of Safety Population.
- The small "n" in summary statistics represents the total number of Patients.
- SD = Standard Deviation, min=minimum, max=maximum
- Programmer Note: Visit x: Visit 2, Visit 5, Visit 7, Visit 9 and Visit 10.
- Source: Listing 16.2.2.2



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.1.3. Summary of Medical and Surgical History (Safety Population)

| System Organ Class /Preferred Term | N = xx |
|-------------------------------------------|------------|
| | n (%) |
| Patient with any medical/Surgical history | xx (xx.xx) |
| System Organ Class 1 | xx (xx.xx) |
| Preferred Term 1 | xx (xx.xx) |
| Preferred Term 2 | xx (xx.xx) |
| System Organ Class 2 | xx (xx.xx) |
| Preferred Term 1 | xx (xx.xx) |
| Preferred Term 2 | xx (xx.xx) |
| System Organ Class 3 | xx (xx.xx) |
| Preferred Term 1 | xx (xx.xx) |
| Preferred Term 2 | xx (xx.xx) |
| System Organ Class 4 | xx (xx.xx) |
| Preferred Term 1 | xx (xx.xx) |
| Preferred Term 2 | xx (xx.xx) |
| System Organ Class 5 | xx (xx.xx) |
| Preferred Term 1 | xx (xx.xx) |
| Preferred Term 2 | xx (xx.xx) |

- The Capital "N" in the column header represents the total number of Safety Population.
- The small "n" in summary statistics represents the total number of Patients.
- Percentages in the "Patient with any medical/Surgical history" rows are based on number of Safety Popluation.
- Percentages in the "System Organ Class" and "Preferred Term" rows are based on number of Patient with any medical history.
- Medical histories were coded using MedDRA Ver24.1
- Source :Listing 16.2.3



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.1.4. Summary of Urine Pregnancy Test (Safety Population)

| | N = xx |
|--------------------------------|------------|
| | n (%) |
| Visit x | |
| Urine pregnancy test performed | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| NA | xx (xx.xx) |
| Result | |
| Positive | xx (xx.xx) |
| Negative | xx (xx.xx) |

- The Capital "N" in the column header represents the total number of Safety Population.
- The small "n" in summary statistics represents the total number of Patients.
- Percentage in the "Urine pregnancy test performed" rows are based on the number of Safety Population.
- Percentage in the "Result" rows are based on the number of Patients with Urine Pregnancy test performed.
- SD = Standard Deviation, min=minimum, max=maximum
- Visit x: Visit 1, Visit 2, Visit 5, Visit 7, Visit 9, Visit 10
- Source :Listing 16.2.4.



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.1.5. Summary of IP Medication Accountability (Safety Population)

| | N=xx |
|----------------------------------------------------|----------------|
| Visit x | |
| No. of Dose missed in the treatment period | |
| N | xx |
| Missing | xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | XX.X |
| (min, max) | (xx.xx, xx.xx) |
| No. of Tablets lost in the treatment period | |
| N | xx |
| Missing | xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |
| No. of Tablets returned | |
| N | xx |
| Missing | xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |
| No. of Tablets to be taken in the treatment period | |
| N | xx |
| Missing | xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |
| No. of Tablets consumed in the treatment period | |
| N | xx |
| Missing | xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |
| Compliance (%) | |
| N | xx |
| Missing | xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |

- The Capital "N" in the column header represents the total number of Safety Population.
- The small "n" in summary statistics represents the total number of Patients.
- SD = Standard Deviation, min=minimum, max=maximum.
- Visit x: Visit 5, Visit 7, Visit 9 and Visit 10.
- Source :Listing 16.2.5.1 and Listing 16.2.5.2



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.2.1. Analysis of change in HbA1c from baseline to Week 24 (Safety Population)

| | Observed value<br>(N = xx) | Change from Baseline<br>(N = xx) | % Change from Baseline<br>(N = xx) |
|---|---|---|---|
| Baseline (Visit 2) | | | |
| N | xxx | | |
| Missing | xx | | |
| Mean (SD) | xx.x (xx.xx) | | |
| Median | xx.x | | |
| (min, max) | (xx.xx, xx.xx) | | |
| Week 24 | | | |
| N | Xx | Xx | xx |
| Missing | Xx | Xx | Xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x |
| (min, max) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| p-value | | x.xxx | x.xxx |

- The Capital "N" in the column header represents the total number of Patients in Safety Population.
- The small "n" in summary statistics represents the total number of Patients.
- SD = Standard deviation, min=minimum, max=maximum
- Change from Baseline Post-Baseline Baseline
- % Change from Baseline = (Post-Baseline Baseline / Baseline) X 100
- p-value calculate using Paired t test / Wilcoxon signed-rank test.
- Source : Listing 16.2.6.1



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.2.2. Analysis of change in Weight from baseline to Week 24. (Safety Population)

| | Observed value<br>(N = xx) | Change from Baseline<br>(N = xx) | % Change from Baseline<br>(N = xx) |
|---|---|---|---|
| Baseline (Visit 2) | (c. im, | ( | (1.1 1.1.1) |
| N | xx | | |
| Missing | xx | | |
| Mean (SD) | xx.x (xx.xx) | | |
| Median | xx.x | | |
| (min, max) | (xx.xx, xx.xx) | | |
| Week 24 | , , | | |
| N | Xx | Xx | xx |
| Missing | Xx | Xx | Xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | xx.x |
| (min, max) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| p-value | | x.xxx | x.xxx |

- The Capital "N" in the column header represents the total number of Patients in Safety Population.
- The small "n" in summary statistics represents the total number of Patients.
- SD = Standard deviation, min=minimum, max=maximum
- Change from Baseline Post-Baseline Baseline
- % Change from Baseline = (Post-Baseline Baseline / Baseline) X 100
- p-value calculate using Paired t test / Wilcoxon signed-rank test.
- Source : Listing 16.2.2.2



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.2.3. Analysis of change in Blood Pressure from baseline to Week 24. (Safety Population)

| | Observed value | Change from Baseline | % Change from Baseline |
|---|---|---|---|
| | (N = xx) | (N = xx) | (N = xx) |
| Systolic Blood Pressure | | | |
| Baseline (Visit 2) | | | |
| N | xx | | |
| Missing | xx | | |
| Mean (SD) | xx.x (xx.xx) | | |
| Median | xx.x | | |
| (min, max) | (xx.xx, xx.xx) | | |
| Week 24 | | | |
| N | xx | XX | xx |
| Missing | xx | xx | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | XX.X | xx.x |
| (min, max) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| p-value | | x.xxx | x.xxx |
| Diastolic Blood Pressure | | | |
| Baseline (Visit 2) | | | |
| N | xx | | |
| Missing | xx | | |
| Mean (SD) | xx.x (xx.xx) | | |
| Median | xx.x | | |
| (min, max) | (xx.xx, xx.xx) | | |
| Week 24 | | | |
| N | xx | xx | xx |
| Missing | xx | XX | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | XX.X | xx.x |
| (min, max) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| p-value | | x.xxx | x.xxx |

- The Capital "N" in the column header represents the total number of Patients in Safety Population.
- The small "n" in summary statistics represents the total number of Patients.
- SD = Standard deviation, min=minimum, max=maximum
- Change from Baseline Post-Baseline Baseline
- % Change from Baseline = (Post-Baseline Baseline / Baseline) X 100
- p-value calculate using Paired t test / Wilcoxon signed-rank test.
- Source : Listing 16.3.5



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.2.4. Analysis of change in Fasting Plasma Glucose from baseline to Week 24. (Safety Population)

| | Observed value<br>(N = xx) | Change from Baseline<br>(N = xx) | % Change from Baseline<br>(N = xx) |
|---|---|---|---|
| Baseline (Visit 2) | • | • | • |
| N | xx | | |
| Missing | xx | | |
| Mean (SD) | xx.x (xx.xx) | | |
| Median | xx.x | | |
| (min, max) | (xx.xx, xx.xx) | | |
| Week 24 | | | |
| N | Xx | Xx | xx |
| Missing | Xx | Xx | Xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x |
| (min, max) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| p-value | | x.xxx | x.xxx |

- The Capital "N" in the column header represents the total number of Patients in Safety Population.
- The small "n" in summary statistics represents the total number of Patients.
- SD = Standard deviation, min=minimum, max=maximum
- Change from Baseline = Post-Baseline Baseline
- % Change from Baseline = (Post-Baseline Baseline / Baseline) X 100
- p-value calculate using paired t test.
- Source : Listing 16.2.6.1



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.2.5. Summary of HbA1c and Fasting Plasma Glucose (Safety Population)

| | N=xx |
|--------------------------------------------------|----------------|
| Visit 1 | |
| HbA1c (%) | |
| N | xx |
| Missing | xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |
| Duration of Type 2 Diabetes Mellitus (in months) | |
| N | xx |
| Missing | XX |
| Mean (SD) | xx.x (xx.xx) |
| Median | XX.X |
| (min, max) | (xx.xx, xx.xx) |
| Visit x | |
| HbA1c and Fasting Plasma Glucose assessed | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| HbA1c (%) | |
| N | xx |
| Missing | xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |
| Fasting Plasma Glucose (mg/dL) | |
| N | xx |
| Missing | xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |

- The Capital "N" in the column header represents the total number of Safety Population.
- The small "n" in summary statistics represents the total number of Patients.
- Percentage in the "HbA1c and Fasting Plasma Glucose Assessed" rows are based on the number of Safety Population.
- SD = Standard Deviation, min=minimum, max=maximum
- Visit x: Visit 2, Visit 5, Visit 7, Visit 9 and Visit 10
- Source :Listing 16.2.6.1



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.3.5. Summary of Hypoglycemic Event (Safety Population).

| | N = xx |
|----------------------------------------------------|----------------|
| | n (%) |
| Patient Experience any hypoglycemic event | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| Event occur Time | |
| Sleeping Time | xx (xx.xx) |
| Day Time | xx (xx.xx) |
| Other Time | xx (xx.xx) |
| Symptoms are present | the feature of |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| Symptoms are present, If Yes | , |
| An irregular heart rhythm | xx (xx.xx) |
| Fatigue | xx (xx.xx) |
| Pale skin | xx (xx.xx) |
| Shakiness | xx (xx.xx) |
| Anxiety | xx (xx.xx) |
| Sweating | xx (xx.xx) |
| Hunger | xx (xx.xx) |
| Irritability | xx (xx.xx) |
| Tingling sensation around the mouth | xx (xx.xx) |
| Crying out during sleep | xx (xx.xx) |
| Other | xx (xx.xx) |
| Possible contributing factors of the event | ^^ (^^.^^) |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| Possible contributing factors of the event, If Yes | ^^ (^^.^^) |
| Alcohol consumption | xx (xx.xx) |
| Concurrent illness | xx (xx.xx) |
| Overdose of IP/Deviation from dosin | xx (xx.xx) |
| Physical Activity | |
| Other | xx (xx.xx) |
| | xx (xx.xx) |
| Fingerstick value obtained at the time of event | () |
| Yes<br>No | xx (xx.xx) |
| | xx (xx.xx) |
| Plasma glucose (mg/dL) | V |
| n<br>Mississa | Xx |
| Missing | Xx |
| Mean (SD)<br>Median | xx.x (xx.xx) |
| 1112 | XX.X |
| (min, max) | (xx.xx, xx.xx) |
| Glucose (mg/dL) | V |
| N<br>Missing | Xx |
| Missing Many (CD) | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | XX.X |
| (min, max) | (xx.xx, xx.xx) |
| Treatment intervention needed for recovery Yes | xx (xx.xx) |
| Document | Page 29 of 71 |
| op ctar y and community bounders | 1 460 23 01 71 |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

| No | xx (xx.xx) |
|---|---|
| Episode treated | , , |
| Drink/Food | xx (xx.xx) |
| Glucose Injection | xx (xx.xx) |
| Other | xx (xx.xx) |
| Indicate assistance needed | |
| None – Subject treated self | xx (xx.xx) |
| Patient was capable of treating self, but received assistance | xx (xx.xx) |
| Patient was not capable of treating self and received assistance | xx (xx.xx) |
| Patient recover post treatment | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |

- The Capital "N" in the column header represents the total number of Safety Population.
- The small "n" in summary statistics represents the total number of Patients.
- Percentages in the "Patient Experience any hypoglycemic event" rows are based on the number of Safety Population.
- Percentages in the "Event occur Time, Symptoms are present, Possible contributing factors of the event, Fingerstick value obtained at the time of event, Treatment intervention needed for recovery, Episode treated, Indicate assistance needed, Patient recover post treatment" rows are based on Patient Experience any hypoglycemic event.
- Percentages in the "Symptoms are present, If Yes" rows are based on Patient Symptoms are present.
- Percentages in the "Possible contributing factors of the event, If Yes" rows are based on Patient Possible contributing factors of the event.
- SD = Standard Deviation, min=minimum, max=maximum
- Source :Listing 16.2.7.1 and Listing 16.2.7.2



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.3.1. Summary of Adverse Event (Safety Population)

| Patient experience any Adverse Event xx (xx.xx) Yes xx (xx.xx) No xx (xx.xx) Relationship xx (xx.xx) Certain xx (xx.xx) Probable/likely xx (xx.xx) Opasible xx (xx.xx) Unlikely xx (xx.xx) Action taken xx (xx.xx) None xx (xx.xx) Change in the study drug administration xx (xx.xx) Drug Withdrawn xx (xx.xx) Dose reduced xx (xx.xx) Dose increased xx (xx.xx) Dose increased xx (xx.xx) Drug treatment required xx (xx.xx) Non-drug treatment required xx (xx.xx) Hospitalization/prolonged hospitalization xx (xx.xx) Diagnostic or clinical test(s) conducted xx (xx.xx) Patient discontinued from the study xx (xx.xx) Severity xx (xx.xx) Mild xx (xx.xx) Moderate xx (xx.xx) Severe xx (xx.xx) Outcome xx (xx.xx) <th< th=""><th></th><th>N = xx</th></th<> | | N = xx |
|---|---|---|
| Yes XX (XXXX) NO XX (XXXX) Relationship XX (XXXXX) Probable/Likely XX (XXXXX) Possible XX (XXXXX) Not related XX (XXXXX) Action taken XX (XXXXX) None XX (XXXXX) Change in the study drug administration XX (XXXXX) Drug Withdrawn XX (XXXXX) Dose reduced XX (XXXXX) Dose increased XX (XXXXX) Dose increased XX (XXXXX) Drug treatment required XX (XXXXX) Non-drug treatment required XX (XXXXX) Hospitalization/prolonged hospitalization XX (XXXXX) Diagnostic or clinical test(s) conducted XX (XXXXX) Patient discontinued from the study XX (XXXXX) Severity XX (XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | n (%) |
| No xx (xx.xx) Relationship xx (xx.xx) Probable/Likely xx (xx.xx) Possible xx (xx.xx) Unlikely xx (xx.xx) Not related xx (xx.xx) Action taken xx (xx.xx) Change in the study drug administration xx (xx.xx) Drug withdrawn xx (xx.xx) Drug interrupted xx (xx.xx) Dose reduced xx (xx.xx) Dose reduced xx (xx.xx) Dose increased xx (xx.xx) Dose increased xx (xx.xx) Dose increased xx (xx.xx) Hospitalization/prolonged hospitalization xx (xx.xx) Diagnostic or clinical test(s) conducted xx (xx.xx) Patient discontinued from the study xx (xx.xx) Severity xx (xx.xx) Wild xx (xx.xx) Severity xx (xx.xx) Wild xx (xx.xx) Severed xx (xx.xx) Severed without sequelae xx (xx.xx) Recovered with sequelae xx (xx.xx) R | Patient experience any Adverse Event | |
| Relationship xx (xx,xx) Certain xx (xx,xx) Probable/Likely xx (xx,xx) Possible xx (xx,xx) Unlikely xx (xx,xx) Not related xx (xx,xx) Action taken xx (xx,xx) None xx (xx,xx) Change in the study drug administration xx (xx,xx) Drug Withdrawn xx (xx,xx) Drug miterrupted xx (xx,xx) Dose reduced xx (xx,xx) Dose increased xx (xx,xx) Drug treatment required xx (xx,xx) Won-drug treatment required xx (xx,xx) Hospitalization/prolonged hospitalization xx (xx,xx) Diagnostic or clinical test(s) conducted xx (xx,xx) Patient discontinued from the study xx (xx,xx) Severety xx (xx,xx) Will xx (xx,xx) Moderate xx (xx,xx) Severe xx (xx,xx) Outcome xx (xx,xx) Recovered without sequelae xx (xx,xx) Not recovered/y Not resolved xx (xx,xx) | Yes | xx (xx.xx) |
| Certain xx (xx.xx) Probable/Likely xx (xx.xx) Possible xx (xx.xx) Unlikely xx (xx.xx) Nor elated xx (xx.xx) Action taken xx (xx.xx) None xx (xx.xx) Change in the study drug administration xx (xx.xx) Drug Withdrawn xx (xx.xx) Drug treatment required xx (xx.xx) Dose increased xx (xx.xx) Dose increased xx (xx.xx) Drug treatment required xx (xx.xx) Hospitalization/prolonged hospitalization xx (xx.xx) Diagnostic or clinical test(s) conducted xx (xx.xx) Patient discontinued from the study xx (xx.xx) Severity xx (xx.xx) Mild xx (xx.xx) Severer xx (xx.xx) Outcome xx (xx.xx) Recovered without sequelae xx (xx.xx) Recovered with sequelae xx (xx.xx) Recovered with sequelae xx (xx.xx) Not recovered/ Not resolved xx (xx.xx) Recovered with sequelae | No | xx (xx.xx) |
| Probable/Likely xx (xx.xx) Possible xx (xx.xx) Unlikely xx (xx.xx) Not related xx (xx.xx) Action taken xx (xx.xx) None xx (xx.xx) Change in the study drug administration xx (xx.xx) Drug Withdrawn xx (xx.xx) Drug interrupted xx (xx.xx) Dose reduced xx (xx.xx) Dose increased xx (xx.xx) Drug treatment required xx (xx.xx) Non-drug treatment required xx (xx.xx) Hospitalization/prolonged hospitalization xx (xx.xx) Patient discontinued from the study xx (xx.xx) Patient discontinued from the study xx (xx.xx) Severity xx (xx.xx) Mild xx (xx.xx) Moderate xx (xx.xx) Severe xx (xx.xx) Outcome xx (xx.xx) Recovered without sequelae xx (xx.xx) Recovered with sequelae xx (xx.xx) Recovering/ resolving xx (xx.xx) Unknown xx (xx.xx) < | Relationship | |
| Possible xx (xx,xx) Unlikely xx (xx,xx) Not related xx (xx,xx) Action taken xx (xx,xx) None xx (xx,xx) Change in the study drug administration xx (xx,xx) Drug Withdrawn xx (xx,xx) Dose increased xx (xx,xx) Dose reduced xx (xx,xx) Dose increased xx (xx,xx) Non-drug treatment required xx (xx,xx) Non-drug treatment required xx (xx,xx) Non-drug treatment required xx (xx,xx) Hospitalization/prolonged hospitalization xx (xx,xx) Diagnostic or clinical test(s) conducted xx (xx,xx) Patient discontinued from the study xx (xx,xx) Severity xx (xx,xx) Mild xx (xx,xx) Moderate xx (xx,xx) Severe xx (xx,xx) Outcome xx (xx,xx) Recovered with sequelae xx (xx,xx) Recovered with sequelae xx (xx,xx) Not recovered/ Not resolved xx (xx,xx) Recovering/ resolving <td>Certain</td> <td>xx (xx.xx)</td> | Certain | xx (xx.xx) |
| Unlikely | Probable/Likely | xx (xx.xx) |
| Unlikely xx (xx.xx) Not related xx (xx.xx) Action taken xx (xx.xx) None xx (xx.xx) Change in the study drug administration xx (xx.xx) Drug Withdrawn xx (xx.xx) Drug treatment required xx (xx.xx) Dose increased xx (xx.xx) Dose increased xx (xx.xx) Drug treatment required xx (xx.xx) Hospitalization/prolonged hospitalization xx (xx.xx) Hospitalization/prolonged hospitalization xx (xx.xx) Diagnostic or clinical test(s) conducted xx (xx.xx) Patient discontinued from the study xx (xx.xx) Severity xx (xx.xx) Mild xx (xx.xx) Moderate xx (xx.xx) Severe xx (xx.xx) Outcome xx (xx.xx) Recovered with sequelae xx (xx.xx) Not recovered hoth resolved xx (xx.xx) Recovering/ resolving xx (xx.xx) Unknown xx (xx.xx) Fatal xx (xx.xx) No xx (xx.x | Possible | xx (xx.xx) |
| Not related xx (xx.xx) Action taken xx (xx.xx) None xx (xx.xx) Change in the study drug administration xx (xx.xx) Drug Withdrawn xx (xx.xx) Drug interrupted xx (xx.xx) Dose reduced xx (xx.xx) Dose increased xx (xx.xx) Drug treatment required xx (xx.xx) Non-drug treatment required xx (xx.xx) Hospitalization/prolonged hospitalization xx (xx.xx) Patient discontinued from the study xx (xx.xx) Severity xx (xx.xx) Mild xx (xx.xx) Moderate xx (xx.xx) Severe xx (xx.xx) Outcome xx (xx.xx) Recovered without sequelae xx (xx.xx) Recovered with sequelae xx (xx.xx) Not recovered/ Not resolved xx (xx.xx) Recovering/ resolving xx (xx.xx) Unknown xx (xx.xx) Fatal xx (xx.xx) Ves xx (xx.xx) No xx (xx.xx) UnE | Unlikely | • • |
| Action taken xx (xx.xx) None xx (xx.xx) Change in the study drug administration xx (xx.xx) Drug Withdrawn xx (xx.xx) Dose increased xx (xx.xx) Dose increased xx (xx.xx) Drug treatment required xx (xx.xx) Non-drug treatment required xx (xx.xx) Non-drug treatment required xx (xx.xx) Hospitalization/prolonged hospitalization xx (xx.xx) Diagnostic or clinical test(s) conducted xx (xx.xx) Patient discontinued from the study xx (xx.xx) Severity xx (xx.xx) Mild xx (xx.xx) Moderate xx (xx.xx) Severered xx (xx.xx) Outcome xx (xx.xx) Recovered without sequelae xx (xx.xx) Recovered with sequelae xx (xx.xx) Recovered with sequelae xx (xx.xx) Recovering/ resolving xx (xx.xx) Unknown xx (xx.xx) Fatal xx (xx.xx) Fatal xx (xx.xx) No xx (xx. | • | |
| Change in the study drug administration | Action taken | The (contrary) |
| Change in the study drug administration | | xx (xx.xx) |
| Drug Withdrawn xx (xx.xx) Drug interrupted xx (xx.xx) Dose reduced xx (xx.xx) Dose increased xx (xx.xx) Drug treatment required xx (xx.xx) Non-drug treatment required xx (xx.xx) Hospitalization/prolonged hospitalization xx (xx.xx) Diagnostic or clinical test(s) conducted xx (xx.xx) Patient discontinued from the study xx (xx.xx) Severity Will Mild xx (xx.xx) Moderate xx (xx.xx) Severe xx (xx.xx) Outcome xx (xx.xx) Recovered without sequelae xx (xx.xx) Recovered with sequelae xx (xx.xx) Recovering/ resolving xx (xx.xx) Unknown xx (xx.xx) Treatment Taken xx (xx.xx) Yes xx (xx.xx) No xx (xx.xx) UnExpected xx (xx.xx) No xx (xx.xx) UnExpected xx (xx.xx) No xx (xx.xx) UnExpected | | |
| Drug interrupted xx (xx.xx) Dose reduced xx (xx.xx) Dose increased xx (xx.xx) Drug treatment required xx (xx.xx) Non-drug treatment required xx (xx.xx) Hospitalization/prolonged hospitalization xx (xx.xx) Diagnostic or clinical test(s) conducted xx (xx.xx) Patient discontinued from the study xx (xx.xx) Severity xx (xx.xx) Mild xx (xx.xx) Moderate xx (xx.xx) Severe xx (xx.xx) Outcome xx (xx.xx) Recovered without sequelae xx (xx.xx) Not recovered/ Not resolved xx (xx.xx) Not recovered/ Not resolved xx (xx.xx) Recovering/ resolving xx (xx.xx) Unknown xx (xx.xx) Fatal xx (xx.xx) Yes xx (xx.xx) No xx (xx.xx) Expected xx (xx.xx) UnExpected xx (xx.xx) No xx (xx.xx) No xx (xx.xx) SAE | | |
| Dose reduced xx (xx.xx) Dose increased xx (xx.xx) Drug treatment required xx (xx.xx) Non-drug treatment required xx (xx.xx) Hospitalization/prolonged hospitalization xx (xx.xx) Diagnostic or clinical test(s) conducted xx (xx.xx) Patient discontinued from the study xx (xx.xx) Severity wx (xx.xx) Mild xx (xx.xx) Moderate xx (xx.xx) Severe xx (xx.xx) Outcome xx (xx.xx) Recovered without sequelae xx (xx.xx) Recovered with sequelae xx (xx.xx) Not recovered/ Not resolved xx (xx.xx) Recovering/ resolving xx (xx.xx) Unknown xx (xx.xx) Fatal xx (xx.xx) Treatment Taken xx (xx.xx) Yes xx (xx.xx) No xx (xx.xx) Expected xx (xx.xx) UnExpected xx (xx.xx) No xx (xx.xx) Yes xx (xx.xx) No x | _ | |
| Dose increased xx (xx.xx) Drug treatment required xx (xx.xx) Non-drug treatment required xx (xx.xx) Hospitalization/prolonged hospitalization xx (xx.xx) Diagnostic or clinical test(s) conducted xx (xx.xx) Patient discontinued from the study xx (xx.xx) Severity xx (xx.xx) Mild xx (xx.xx) Moderate xx (xx.xx) Severe xx (xx.xx) Outcome xx (xx.xx) Recovered without sequelae xx (xx.xx) Recovered with sequelae xx (xx.xx) Not recovered/ Not resolved xx (xx.xx) Recovering/ resolving xx (xx.xx) Unknown xx (xx.xx) Fatal xx (xx.xx) Treatment Taken xx (xx.xx) Yes xx (xx.xx) No xx (xx.xx) SAE xx (xx.xx) UnExpected xx (xx.xx) No xx (xx.xx) SAE xx (xx.xx) No xx (xx.xx) SAE Criteria xx (xx | | |
| Drug treatment required | | |
| Non-drug treatment required xx (xx.xx) Hospitalization/prolonged hospitalization xx (xx.xx) Diagnostic or clinical test(s) conducted xx (xx.xx) Patient discontinued from the study xx (xx.xx) Severity xx (xx.xx) Mild xx (xx.xx) Moderate xx (xx.xx) Severe xx (xx.xx) Outcome xx (xx.xx) Recovered without sequelae xx (xx.xx) Recovered with sequelae xx (xx.xx) Not recovered/Not resolved xx (xx.xx) Recovering/ resolving xx (xx.xx) Unknown xx (xx.xx) Fatal xx (xx.xx) Treatment Taken xx (xx.xx) Yes xx (xx.xx) No xx (xx.xx) Expected xx (xx.xx) UnExpected xx (xx.xx) SAE xx (xx.xx) No xx (xx.xx) No xx (xx.xx) No xx (xx.xx) SAE Criteria xx (xx.xx) Result in Death in-patient hospitalisation | | |
| Hospitalization/prolonged hospitalization xx (xx.xx) Diagnostic or clinical test(s) conducted xx (xx.xx) Patient discontinued from the study xx (xx.xx) xx (xx.x | | |
| Diagnostic or clinical test(s) conducted xx (xx.xx) Patient discontinued from the study xx (xx.xx) Severity xx (xx.xx) Mild xx (xx.xx) Severe xx (xx.xx) Severe xx (xx.xx) Outcome xx (xx.xx) Recovered without sequelae xx (xx.xx) Recovered with sequelae xx (xx.xx) Not recovered/ Not resolved xx (xx.xx) Recovering/ resolving xx (xx.xx) Unknown xx (xx.xx) Fatal xx (xx.xx) Treatment Taken xx (xx.xx) Yes xx (xx.xx) No xx (xx.xx) UnExpected xx (xx.xx) UnExpected xx (xx.xx) Yes xx (xx.xx) No xx (xx.xx) No xx (xx.xx) SAE Xx (xx.xx) No xx (xx.xx) No xx (xx.xx) No xx (xx.xx) SAE Xx (xx.xx) No xx (xx.xx) | · | |
| Patient discontinued from the study xx (xx.xx) Severity xx (xx.xx) Mild xx (xx.xx) Moderate xx (xx.xx) Severe xx (xx.xx) Outcome xx (xx.xx) Recovered without sequelae xx (xx.xx) Recovered with sequelae xx (xx.xx) Not recovered/ Not resolved xx (xx.xx) Recovering/ resolving xx (xx.xx) Unknown xx (xx.xx) Fatal xx (xx.xx) Yes xx (xx.xx) No xx (xx.xx) Expectedness xx (xx.xx) Expected xx (xx.xx) UnExpected xx (xx.xx) SAE xx (xx.xx) No xx (xx.xx) No xx (xx.xx) SAE xx (xx.xx) No xx (xx.xx) No xx (xx.xx) No xx (xx.xx) No xx (xx.xx) No xx (xx.xx) No xx (xx.xx) No xx (xx.xx) <td></td> <td></td> | | |
| Severity xx (xx.xx) Mild xx (xx.xx) Moderate xx (xx.xx) Severe xx (xx.xx) Outcome xx (xx.xx) Recovered without sequelae xx (xx.xx) Recovering/ resolving xx (xx.xx) Unknown xx (xx.xx) Fatal xx (xx.xx) Teatment Taken xx (xx.xx) Yes xx (xx.xx) No xx (xx.xx) Expectedness xx (xx.xx) Expected xx (xx.xx) UnExpected xx (xx.xx) SAE yes Yes xx (xx.xx) No xx (xx.xx) SAE Criteria xx (xx.xx) Result in Death imediately life-threatening xx (xx.xx) New in-patient hospitalisation xx (xx.xx) Prolonged in-patient hospitalisation xx (xx.xx) | | |
| Mild xx (xx.xx) Moderate xx (xx.xx) Severe xx (xx.xx) Outcome xx (xx.xx) Recovered without sequelae xx (xx.xx) Recovering/ resolving xx (xx.xx) Not recovered/ Not resolved xx (xx.xx) Recovering/ resolving xx (xx.xx) Unknown xx (xx.xx) Fatal xx (xx.xx) Treatment Taken xx (xx.xx) Yes xx (xx.xx) No xx (xx.xx) UnExpected xx (xx.xx) SAE xx (xx.xx) Yes xx (xx.xx) No xx (xx.xx) SAE Criteria xx (xx.xx) Result in Death xx (xx.xx) Immediately life-threatening xx (xx.xx) New in-patient hospitalisation xx (xx.xx) Prolonged in-patient hospitalisation xx (xx.xx) | · | the formal of |
| Moderate xx (xx.xx) Severe xx (xx.xx) Outcome xx (xx.xx) Recovered without sequelae xx (xx.xx) Recovered/ Not resolved xx (xx.xx) Recovering/ resolving xx (xx.xx) Unknown xx (xx.xx) Fatal xx (xx.xx) Fatal xx (xx.xx) Fatal xx (xx.xx) Treatment Taken xx (xx.xx) Yes xx (xx.xx) No xx (xx.xx) Expectedness xx (xx.xx) Expected xx (xx.xx) SAE xx (xx.xx) Yes xx (xx.xx) No xx (xx.xx) SAE Criteria xx (xx.xx) Result in Death xx (xx.xx) immediately life-threatening xx (xx.xx) New in-patient hospitalisation xx (xx.xx) Prolonged in-patient hospitalisation xx (xx.xx) | - | xx (xx.xx) |
| Severe xx (xx.xx) Outcome xx (xx.xx) Recovered without sequelae xx (xx.xx) Recovering with sequelae xx (xx.xx) Not recovered/ Not resolved xx (xx.xx) Recovering/ resolving xx (xx.xx) Unknown xx (xx.xx) Fatal xx (xx.xx) Fatal xx (xx.xx) Yes xx (xx.xx) No xx (xx.xx) Expectedness xx (xx.xx) Expected xx (xx.xx) UnExpected xx (xx.xx) SAE xx (xx.xx) Yes xx (xx.xx) No xx (xx.xx) SAE Criteria xx (xx.xx) Result in Death xx (xx.xx) immediately life-threatening xx (xx.xx) New in-patient hospitalisation xx (xx.xx) Prolonged in-patient hospitalisation xx (xx.xx) | | |
| Outcome Recovered without sequelae xx (xx.xx) Recovered/ Not resolved xx (xx.xx) Not recovering/ resolving xx (xx.xx) Unknown xx (xx.xx) Fatal xx (xx.xx) Treatment Taken xx (xx.xx) Yes xx (xx.xx) No xx (xx.xx) Expectedness xx (xx.xx) Expected xx (xx.xx) UnExpected xx (xx.xx) SAE xx (xx.xx) Yes xx (xx.xx) No xx (xx.xx) SAE Criteria xx (xx.xx) Result in Death in Death immediately life-threatening xx (xx.xx) xx (xx.xx) New in-patient hospitalisation xx (xx.xx) xx (xx.xx) Prolonged in-patient hospitalisation xx (xx.xx) xx (xx.xx) | Severe | |
| Recovered with sequelae xx (xx.xx) Not recovered/ Not resolved xx (xx.xx) Recovering/ resolving xx (xx.xx) Unknown xx (xx.xx) Fatal xx (xx.xx) Treatment Taken Yes xx (xx.xx) No xx (xx.xx) Expectedness xx (xx.xx) Expected xx (xx.xx) UnExpected xx (xx.xx) SAE xx (xx.xx) Yes xx (xx.xx) No xx (xx.xx) SAE Criteria xx (xx.xx) Result in Death immediately life-threatening xx (xx.xx) xx (xx.xx) New in-patient hospitalisation xx (xx.xx) xx (xx.xx) | | tas (camas) |
| Recovered with sequelae xx (xx.xx) Not recovered/ Not resolved xx (xx.xx) Recovering/ resolving xx (xx.xx) Unknown xx (xx.xx) Fatal xx (xx.xx) Treatment Taken Yes xx (xx.xx) No xx (xx.xx) Expectedness xx (xx.xx) Expected xx (xx.xx) UnExpected xx (xx.xx) SAE xx (xx.xx) Yes xx (xx.xx) No xx (xx.xx) SAE Criteria xx (xx.xx) Result in Death immediately life-threatening xx (xx.xx) xx (xx.xx) New in-patient hospitalisation xx (xx.xx) xx (xx.xx) | Recovered without sequelae | xx (xx.xx) |
| Not recovered/ Not resolved xx (xx.xx) Recovering/ resolving xx (xx.xx) Unknown xx (xx.xx) Fatal xx (xx.xx) Treatment Taken Yes xx (xx.xx) No xx (xx.xx) Expectedness xx (xx.xx) Expected xx (xx.xx) UnExpected xx (xx.xx) SAE xx (xx.xx) Yes xx (xx.xx) No xx (xx.xx) SAE Criteria xx (xx.xx) Result in Death xx (xx.xx) immediately life-threatening xx (xx.xx) New in-patient hospitalisation xx (xx.xx) Prolonged in-patient hospitalisation xx (xx.xx) | | |
| Recovering/ resolving | · | |
| Unknown xx (xx.xx) Fatal xx (xx.xx) Treatment Taken xx (xx.xx) Yes xx (xx.xx) No xx (xx.xx) Expectedness xx (xx.xx) UnExpected xx (xx.xx) SAE xx (xx.xx) Yes xx (xx.xx) No xx (xx.xx) SAE Criteria xx (xx.xx) Result in Death xx (xx.xx) immediately life-threatening xx (xx.xx) New in-patient hospitalisation xx (xx.xx) Prolonged in-patient hospitalisation xx (xx.xx) | | the state of the s |
| Fatal xx (xx.xx) Treatment Taken xx (xx.xx) Yes xx (xx.xx) No xx (xx.xx) Expectedness xx (xx.xx) UnExpected xx (xx.xx) SAE xx (xx.xx) Yes xx (xx.xx) No xx (xx.xx) SAE Criteria xx (xx.xx) Result in Death immediately life-threatening immediately life-threatening immediately life-threatening important hospitalisation important hospitalisation important hospitalisation important hospitalisation important | | |
| Treatment Taken xx (xx.xx) Yes xx (xx.xx) No xx (xx.xx) Expectedness xx (xx.xx) UnExpected xx (xx.xx) SAE xx (xx.xx) Yes xx (xx.xx) No xx (xx.xx) SAE Criteria xx (xx.xx) Result in Death immediately life-threatening immediately life-threateni | Fatal | |
| No xx (xx.xx) Expectedness Expected xx (xx.xx) UnExpected xx (xx.xx) SAE Yes xx (xx.xx) No xx (xx.xx) SAE Criteria Result in Death xx (xx.xx) immediately life-threatening xx (xx.xx) New in-patient hospitalisation xx (xx.xx) Prolonged in-patient hospitalisation xx (xx.xx) | Treatment Taken | , , |
| No xx (xx.xx) Expectedness Expected xx (xx.xx) UnExpected xx (xx.xx) SAE Yes xx (xx.xx) No xx (xx.xx) SAE Criteria Result in Death xx (xx.xx) immediately life-threatening xx (xx.xx) New in-patient hospitalisation xx (xx.xx) Prolonged in-patient hospitalisation xx (xx.xx) | Yes | xx (xx.xx) |
| Expected xx (xx.xx) UnExpected xx (xx.xx) SAE Yes xx (xx.xx) No xx (xx.xx) SAE Criteria Result in Death xx (xx.xx) immediately life-threatening xx (xx.xx) New in-patient hospitalisation xx (xx.xx) Prolonged in-patient hospitalisation xx (xx.xx) | No | |
| Expected xx (xx.xx) UnExpected xx (xx.xx) SAE Yes xx (xx.xx) No xx (xx.xx) SAE Criteria Result in Death xx (xx.xx) immediately life-threatening xx (xx.xx) New in-patient hospitalisation xx (xx.xx) Prolonged in-patient hospitalisation xx (xx.xx) | Expectedness | |
| Yes xx (xx.xx) No xx (xx.xx) SAE Criteria Result in Death xx (xx.xx) immediately life-threatening xx (xx.xx) New in-patient hospitalisation xx (xx.xx) Prolonged in-patient hospitalisation xx (xx.xx) | | xx (xx.xx) |
| Yes xx (xx.xx) No xx (xx.xx) SAE Criteria Result in Death xx (xx.xx) immediately life-threatening xx (xx.xx) New in-patient hospitalisation xx (xx.xx) Prolonged in-patient hospitalisation xx (xx.xx) | UnExpected | xx (xx.xx) |
| No | SAE | |
| SAE Criteria Result in Death immediately life-threatening New in-patient hospitalisation Prolonged in-patient hospitalisation xx (xx.xx) xx (xx.xx) xx (xx.xx) | Yes | xx (xx.xx) |
| Result in Deathxx (xx.xx)immediately life-threateningxx (xx.xx)New in-patient hospitalisationxx (xx.xx)Prolonged in-patient hospitalisationxx (xx.xx) | No | xx (xx.xx) |
| immediately life-threatening xx (xx.xx) New in-patient hospitalisation xx (xx.xx) Prolonged in-patient hospitalisation xx (xx.xx) | SAE Criteria | |
| immediately life-threateningxx (xx.xx)New in-patient hospitalisationxx (xx.xx)Prolonged in-patient hospitalisationxx (xx.xx) | Result in Death | xx (xx.xx) |
| Prolonged in-patient hospitalisation xx (xx.xx) | immediately life-threatening | |
| | New in-patient hospitalisation | xx (xx.xx) |
| Persistent or significant disability/incapacity xx (xx.xx) | Prolonged in-patient hospitalisation | xx (xx.xx) |
| | Persistent or significant disability/incapacity | xx (xx.xx) |
| Document Page 31 o | Document | Page 31 of 71 |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

| Congenital anomaly | xx (xx.xx) |
|--------------------|------------|
| Any Other | xx (xx.xx) |

- The Capital "N" in the column header represents the total number of Safety Population.
- The small "n" in summary statistics represents the total number of Patients.
- Percentages in the "Patient experience any Adverse Event" rows are based on the number of safety Population.
- Percentages in the "Relationship, Action taken, Severity, Outcome, Treatment Taken, Expectedness and SAE" rows are based on the number of Patient experience any Adverse Event.
- Percentage in the "SAE Criteria" rows are based on the number of Patient any SAE.
- Source :Listing 16.3.1.1



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.3.2. Summary of Adverse Event of special interest (Safety Population)

| | N = xx |
|-----------------------------------|------------|
| | n (%) |
| Hypoglycemic Events | xx (xx.xx) |
| Urinary Tract Infection | xx (xx.xx) |
| Gentital Tract Infection | xx (xx.xx) |
| Volume depletion | xx (xx.xx) |
| Diabetic Ketoacidosis | xx (xx.xx) |
| Renal Events | xx (xx.xx) |
| Hospitalization for Heart Failure | xx (xx.xx) |

- The Capital "N" in the column header represents the total number of Safety Population.
- The small "n" in summary statistics represents the total number of Patients.
- Percentages rows are based on the number of safety Population.
- Source :Listing 16.3.7



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.3.3. Summary of Haematology Parameter (Safety Population)

| | N = xx |
|-------------------------|----------------|
| Visit x | |
| Blood Sample Collected | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| Haematology Parameter x | |
| N | Xx |
| Missing | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |

- The Capital "N" in the column header represents the total number of Safety Population.
- The small "n" in summary statistics represents the total number of Patients.
- SD = Standard Deviation, min=minimum, max=maximum;
- Percentages in the "Blood Sample Collected" rows are based on the number of Safety Population.
- Programmer Note: Haematology Parameter x: Hematocrit (%), Leukocyte count (/μL), Neutrophils (%), Basophils (%), Lymphocytes (%), Eosinophils (%), Monocytes (%), Platelet count (/μL), Haemoglobin (g/dL)
- Visit x: Visit 1, Visit 2, Visit 5, Visit 7, Visit 9 and Visit 10
- Source :Listing 16.3.3.1



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.3.4. Summary of Clinical Chemistry Parameter (Safety Population)

| | N = xx |
|--------------------------------|----------------|
| Visit x | |
| Blood Sample Collected | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| Clinical chemistry Parameter x | |
| N | XX |
| Missing | XX |
| Mean (SD) | xx.x (xx.xx) |
| Median | XX.X |
| (min, max) | (xx.xx, xx.xx) |

- The Capital "N" in the column header represents the total number of safety population.
- The small "n" in summary statistics represents the total number of Patients.
- SD = Standard Deviation, min=minimum, max=maximum;
- Percentages in the "Blood Sample Collected" rows are based on the number of Safety Population.
- Programmer Note: Clinical chemistry Parameter x: Creatinine (mg/dL), Total Bilirubin (mg/dL), Alkaline phosphatise (U/L),
   Aspartate transaminase (U/L), Alanine transaminase (U/L), Albumin (g/dL), Potassium (mEq/L), Total Calcium (mg/dL),
   Sodium (mg/dL), Sodium (mmol/L), Sodium (mEq/L) and Creatine kinase (U/L)
- Visit x: Visit 1, Visit 2, Visit 5, Visit 7, Visit 9 and Visit 10
- Source : Listing 16.3.3.2



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.3.5. Summary of Urinalysis (Safety Population)

| | N=xx |
|------------------|------------|
| | n (%) |
| Visit x | |
| Sample collected | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| Blood | |
| Normal | xx (xx.xx) |
| Abnormal NCS | xx (xx.xx) |
| Abnormal CS | xx (xx.xx) |
| Protein | |
| Normal | xx (xx.xx) |
| Abnormal NCS | xx (xx.xx) |
| Abnormal CS | xx (xx.xx) |
| Glucose | |
| Normal | xx (xx.xx) |
| Abnormal NCS | xx (xx.xx) |
| Abnormal CS | xx (xx.xx) |

- The Capital "N" in the column header represents the total number of Safety Population.
- The small "n" in summary statistics represents the total number of Patients.
- Percentages in the "Sample Collected" rows are based on the number of Safety Population.
- Percentages in the "Blood, Protein, Glucose" rows are based on the number of Patient sample collected.
- Visit x: Visit 1, Visit 2, Visit 5, Visit 7, Visit 9 and Visit 10.
- Source : Listing 16.3.3.3


| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.3.6. Summary of Electrocardiogram (Safety Population)

| | (N = xx) |
|------------------------|----------------|
| Visit x | |
| ECG Performed | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| Heart rate (beats/min) | |
| N | xx |
| Missing | XX |
| Mean (SD) | xx.x (xx.xx) |
| Median | XX.X |
| (min, max) | (xx.xx, xx.xx) |
| QRS (ms) | |
| N | XX |
| Missing | XX |
| Mean (SD) | xx.x (xx.xx) |
| Median | XX.X |
| (min, max) | (xx.xx, xx.xx) |
| PR (ms) | • • • |
| N | XX |
| Missing | XX |
| Mean (SD) | xx.x (xx.xx) |
| Median | XX.X |
| (min, max) | (xx.xx, xx.xx) |
| RR (ms) | ( ) |
| N | XX |
| Missing | XX |
| Mean (SD) | xx.x (xx.xx) |
| Median | XX.X |
| (min, max) | (xx.xx, xx.xx) |
| QT (ms) | (y |
| N | XX |
| Missing | XX |
| Mean (SD) | xx.x (xx.xx) |
| Median | XX.X |
| (min, max) | (xx.xx, xx.xx) |
| QTcF (ms) | , , , |
| N | XX |
| Missing | XX |
| Mean (SD) | xx.x (xx.xx) |
| Median | XX.X |
| (min, max) | (xx.xx, xx.xx) |

- The Capital "N" in the column header represents the total number of Safety Population.
- The small "n" in summary statistics represents the total number of Patients.
- SD = Standard Deviation, min=minimum, max=maximum.
- Visit x: Visit 2, Visit 7, Visit 9 and Visit 10
- Source :Listing 16.3.4



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.3.7. Summary of Vital Signs (Safety Population)

| | N = xx |
|---------------------------------|----------------|
| Visit x | |
| Vital Signs Collected | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| Pulse rate (beats/min) | |
| N | XX |
| Missing | XX |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |
| Systolic Blood Pressure (mmHg) | |
| N | Xx |
| Missing | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | XX.X |
| (min, max) | (xx.xx, xx.xx) |
| Diastolic Blood Pressure (mmHg) | , |
| N | XX |
| Missing | xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |
| Respiratory Rate (breaths/min) | , |
| N | Xx |
| Missing | Xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | xx.x |
| (min, max) | (xx.xx, xx.xx) |
| Body Temperature (°F) | (, |
| N | XX |
| Missing | xx |
| Mean (SD) | xx.x (xx.xx) |
| Median | XX.X |
| (min, max) | (xx.xx, xx.xx) |

- The Capital "N" in the column header represents the total number of Safety Population.
- The small "n" in summary statistics represents the total number of Patients.
- Percentage in the "Vital Signs collected" rows are based on the number of Safety Population.
- SD = Standard Deviation, min=minimum, max=maximum;
- Visit x: Visit 1, Visit 2, Visit 5, Visit 7, Visit 9 and Visit 10
- Source : Listing 16.3.5



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.3.8. Summary of Physical examination

| | N = xx |
|--------------------------------|------------|
| | n (%) |
| Visit x | |
| Physical examination performed | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| System x | |
| Normal | xx (xx.xx) |
| Abnormal NCS | xx (xx.xx) |
| Abnormal CS | xx (xx.xx) |

- The Capital "N" in the column header represents the total number Safety Population.
- The small "n" in summary statistics represents the total number of Patients.
- Percentages in the "Physical Examination performed" rows are based on Total number of Patient Safety Population.
- Percentages in the "System x" rows are based on number of Patient Physical Examination performed.
- Programmer Note: Generate summaries for the following System x: General Appearance, Cardiovascular System, Lungs, Abdomen, Extremities, Head Eye Ear Nose Throat (HEENT), Neurological System, Dermatological System, Genito-urinary System and Other.
- NCS= Non-clinically significant
- CS= clinically significant
- Programme Note: Visit 1, Visit 2, Visit 5, Visit 7, Visit 9 and Visit 10
- Source :Listing 16.3.6



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

# Listing 16.2.1.1. Listing of Patients Informed Consent Details

| | Written Informed consent | Date of Written Informed | Time of Written Informed |
|---|---|---|---|
| Patient Number | obtained | Consent Consent | |
| XX-XXX | Yes/No | DD-MMM-YYYY | HH:MM |
| XX-XXX | Yes/No | DD-MMM-YYYY | HH:MM |
| XX-XXX | Yes/No | DD-MMM-YYYY | HH:MM |
| XX-XXX | Yes/No | DD-MMM-YYYY | HH:MM |
| XX-XXX | Yes/No | DD-MMM-YYYY | HH:MM |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

# Listing 16.2.1.2. Listing of Patients End of Treatment

| Patient | | Treatment with study Drug | Date of Last | Most appropriate reason for | Date of Last |
|---|---|---|---|---|---|
| Number | Visit | Discontinued prematurely | Dose taken | withdrawal/Discontinued of Study | contact |
| XX-XXX | XXXX | Yes/No | DD-MMM-YYYY | xxxx | DD-MMM-YYYY |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

# Listing 16.2.1.3. Listing of Patients Study Completion

| Patient | | Patient complete | Date of Completion/ | Primary reason | Other, |
|---|---|---|---|---|---|
| Number | Visit | the study | Discontinuation | for withdrawal | Specify |
| XX-XXX | XXXX | Yes/No | DD-MMM-YYYY | XXXX | xxxx |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## Listing 16.2.1.4. Listing of Analysis Population

| Patient Number | Enrolled Population | Safety Population |
|----------------|---------------------|-------------------|
| xx-xxx | Yes/No | Yes/No |
| xx-xxx | Yes/No | Yes/No |
| xx-xxx | Yes/No | Yes/No |
| xx-xxx | Yes/No | Yes/No |
| XX-XXX | Yes/No | Yes/No |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Listing 16.2.2.1. Listing of Patients Demographics

| Patient Number | Date of Birth | Age (Year) | Gender | Race | Other, Specify |
|---|---|---|---|---|---|
| XX-XXX | DD-MMM-YYYY | XX | Male/Female | Race/Other | XXXX |
| XX-XXX | DD-MMM-YYYY | XX | Male/Female | Race/Other | xxxx |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## Listing 16.2.2.2. Listing of Patients Anthropometric Assessment

| Patient Number | Visit | Height (cm) | Weight (Kg) | Waist Circumference (cm) | Body Mass Index (Kg/m2) |
|---|---|---|---|---|---|
| XX-XXX | XXXX | XXX | XXX | xxx | xxx |
| XX-XXX | XXXX | XXX | XXX | xxx | xxx |
| XX-XXX | XXXX | XXX | XXX | xxx | xxx |
| XX-XXX | XXXX | xxx | XXX | xxx | xxx |
| XX-XXX | XXXX | XXX | xxx | xxx | xxx |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Listing 16.2.3. Listing of Patients Medical History

| Patient | Patient have any | Seq. | Medical/Surgical | Preferred | System | | | | Receiving |
|---|---|---|---|---|---|---|---|---|---|
| Number | Medical/Surgical history | No | Description | Term | Organ Class | Start Date | Stop Date | Ongoing | Treatment |
| xx-xxx | Yes/No | XX | XXXX | xxxx | XXXX | DD-MMM-YYYY | DD-MMM-YYYY | XXXX | Yes/No |
| XX-XXX | Yes/No | XX | XXXX | xxxx | XXXX | DD-MMM-YYYY | DD-MMM-YYYY | XXXX | Yes/No |
| XX-XXX | Yes/No | XX | XXXX | XXXX | XXXX | DD-MMM-YYYY | DD-MMM-YYYY | xxxx | Yes/No |
| XX-XXX | Yes/No | XX | XXXX | XXXX | XXXX | DD-MMM-YYYY | DD-MMM-YYYY | xxxx | Yes/No |
| XX-XXX | Yes/No | XX | XXXX | XXXX | XXXX | DD-MMM-YYYY | DD-MMM-YYYY | xxxx | Yes/No |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Listing 16.2.4. Listing of Patients Urine Pregnancy test (Women of child bearing potential)

| Patient | | Urine Pregnancy | If No, Specify | Date and Time of Urine | |
|---|---|---|---|---|---|
| Number | Visit | test performed | Reason | Sample | Result |
| XX-XXX | XXXX | Yes/No/NA | xxxx | DD-MMM-YYYY/HH:MM | Positive/Negative |
| XX-XXX | XXXX | Yes/No/NA | XXXX | DD-MMM-YYYY/HH:MM | Positive/Negative |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## Listing 16.2.5.1. Listing of Patients IP Dispensing

| Patient | | Study Drug | If No, Specify | Number of Tables | Kit | Kit | Kit |
|---|---|---|---|---|---|---|---|
| Number | Visit | dispensed | Reason | dispensed | Number 1 | Number 2 | Number 3 |
| XX-XXX | XXXX | Yes/No/NA | xxxx | XXXX | xxxx | xxxx/NA | xxxx/NA |
| XX-XXX | XXXX | Yes/No/NA | XXXX | XXXX | XXXX | xxxx/NA | xxxx/NA |
| XX-XXX | XXXX | Yes/No/NA | xxxx | XXXX | xxxx | xxxx/NA | xxxx/NA |
| XX-XXX | XXXX | Yes/No/NA | XXXX | XXXX | XXXX | xxxx/NA | xxxx/NA |
| XX-XXX | XXXX | Yes/No/NA | XXXX | XXXX | XXXX | xxxx/NA | xxxx/NA |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Listing 16.2.5.2. Listing of Patients IP Medication Accountability

| Patient<br>Number | Visit | No. of Dose missed<br>in the treatment<br>Period | No. of Tablets lost<br>in the treatment<br>period | No. of<br>Tablets<br>returned | No. of Tablets to<br>be taken in the<br>treatment period | No. of Tablets<br>consumed in the<br>treatment period | Compliance<br>(%) |
|---|---|---|---|---|---|---|---|
| XX-XXX | XXXX | XX | XX | XX | XX | XX | XXX |
| XX-XXX | XXXX | XX | XX | XX | XX | XX | XXX |
| XX-XXX | XXXX | XX | XX | XX | XX | XX | XXX |
| XX-XXX | XXXX | XX | XX | XX | XX | XX | XXX |
| XX-XXX | XXXX | XX | XX | XX | XX | XX | XXX |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## Listing 16.2.6.1. Listing of Patients HbA1c and Fasting Plasma Glucose

| Patient | | HbA1c and Fasting | Date of HbA1c | HbA1c | Duration of Type 2 Diabetes | Fasting Plasma |
|---|---|---|---|---|---|---|
| Number | Visit | Plasma Glucose assessed | Assessment | (%) | Mellitus (in months) | Glucose (mg/dL) |
| XX-XXX | XXXX | Yes/No | DD-MMM-YYYY | XXXX | xxx | XXX |
| XX-XXX | XXXX | Yes/No | DD-MMM-YYYY | XXXX | xxx | XXX |
| XX-XXX | XXXX | Yes/No | DD-MMM-YYYY | XXXX | xxx | XXX |
| XX-XXX | XXXX | Yes/No | DD-MMM-YYYY | XXXX | xxx | Xxx |
| XX-XXX | XXXX | Yes/No | DD-MMM-YYYY | XXXX | xxx | XXX |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## Listing 16.2.6.2. Listing of Patients Fasting Plasma Glucose

| Patient | | Date and Time of self- | Patient fasting for | Fasting Plasma | Repeated Fasting Plasma | Patient scheduled for | Laboratory |
|---|---|---|---|---|---|---|---|
| Number | Visit | monitoring | 8 hours | glucose (mg/dL) | Glucose (mg/dL) | Laboratory FPG within a week | FPG Value |
| XX-XXX | XXXX | DD-MMM-YYYY/HH:MM | Yes/No | XXX | xxx | yes/no | xxx |
| XX-XXX | XXXX | DD-MMM-YYYY/HH:MM | Yes/No | XXX | xxx | yes/no | XXX |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

## Listing 16.2.7.1. Listing of Patients Hypoglycaemic Event (Part I)

| | | Patient experience | | | | | Any Possible | | Fingerstick value | Plasma | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| <b>Patient</b> | | any hypoglycaemic | Start Date/Stop | Event occur | Symptoms | | Contributing factors | | obtained at the | glucose | Glucose |
| Number | Visit | event | Date | Time | Present | If Yes | of the Event | If Yes | time of event | (mg/dL) | Value |
| | | | DD-MMM-YYYY/ | Sleeping Time/ | | | | | | | |
| XX-XXX | XXXX | Yes/No | DD-MMM-YYYY | Day Time/Other | Yes/No | XXXX | Yes/No | XXXX | Yes/No | Xxx | Xxx |
| | | | DD-MMM-YYYY/ | Sleeping Time/ | | | | | | | |
| XX-XXX | XXXX | Yes/No | DD-MMM-YYYY | Day Time/Other | Yes/No | XXXX | Yes/No | XXXX | Yes/No | Xxx | Xxx |
| | | | DD-MMM-YYYY/ | Sleeping Time/ | | | | | | | |
| XX-XXX | XXXX | Yes/No | DD-MMM-YYYY | Day Time/Other | Yes/No | XXXX | Yes/No | XXXX | Yes/No | Xxx | Xxx |
| | | | DD-MMM-YYYY/ | Sleeping Time/ | | | | | | | |
| XX-XXX | XXXX | Yes/No | DD-MMM-YYYY | Day Time/Other | Yes/No | XXXX | Yes/No | XXXX | Yes/No | XXX | xxx |
| | | | DD-MMM-YYYY/ | Sleeping Time/ | | | | | | | |
| XX-XXX | XXXX | Yes/No | DD-MMM-YYYY | Day Time/Other | Yes/No | XXXX | Yes/No | XXXX | Yes/No | XXX | XXX |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## Listing 16.2.7.2. Listing of Patients Hypoglycaemic Event (Part II)

| Patient | | Treatment intervention | How was the Episode | Indicate assistance | Patient recover | Time of last IP | Time of | Meal |
|---|---|---|---|---|---|---|---|---|
| Number | Visit | needed for recovery | treated | needed | post treatment | administration | last meal | content |
| | | | (Drink/Food)/ (Glucose | | | | | |
| XX-XXX | XXXX | Yes/No | Injection)/Other | XXXX | Yes/No | HH:MM | HH:MM | XXXX |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

Listing 16.3.1.1. Listing of Patients Adverse Event Assessment

| Patient Number | Visit | Patient Experience any Adverse Event Since last visit |
|---|---|---|
| XX-XXX | XXXX | Yes/No |
| XX-XXX | XXXX | Yes/No |
| XX-XXX | XXXX | Yes/No |
| XX-XXX | XXXX | Yes/No |
| XX-XXX | XXXX | Yes/No |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Chalistical Analysis Dlan | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

## Listing 16.3.1.2. Listing of Patients Adverse Event

| Patient | Patient Experience | Seq. | Event | Start Date/ End | | Action | | | | Treatment | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Number | Any Adverse Event | No | Description | Date | Ongoing | Relationship | taken | Severity | Outcome | taken | Expectedness | SAE |
| | | | | DD-MMM-YYYY/ | | | | | | | Expected/ | |
| XX-XXX | Yes/No | XX | XXX | DD-MMM-YYYY | XXX | xxx | XXX | XXX | xxx | Yes/No | Unexpected | Yes/No |
| | | | | DD-MMM-YYYY/ | | | | | | | Expected/ | |
| XX-XXX | Yes/No | XX | XXX | DD-MMM-YYYY | XXX | XXX | XXX | XXX | xxx | Yes/No | Unexpected | Yes/No |
| | | | | DD-MMM-YYYY/ | | | | | | | Expected/ | |
| XX-XXX | Yes/No | XX | XXX | DD-MMM-YYYY | XXX | XXX | XXX | XXX | xxx | Yes/No | Unexpected | Yes/No |
| | | | | DD-MMM-YYYY/ | | | | | | | Expected/ | |
| XX-XXX | Yes/No | XX | xxx | DD-MMM-YYYY | XXX | XXX | XXX | XXX | xxx | Yes/No | Unexpected | Yes/No |
| | | | | DD-MMM-YYYY/ | | | | | | | Expected/ | |
| XX-XXX | Yes/No | XX | XXX | DD-MMM-YYYY | XXX | XXX | XXX | XXX | XXX | Yes/No | Unexpected | Yes/No |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## Listing 16.3.2. Listing of Patients Serious Adverse Event

| | | | | | Date Investigator | Patient | | | | | _ |
|---|---|---|---|---|---|---|---|---|---|---|---|
| <b>Patient</b> | | | SAE | Date of AE met | became aware of | hospitalised | Date of | Date of | Seriousness | Date of Event | Outcome |
| Number | Age | Gender | Term | criteria for SAE | serious AE | due to SAE | Hospitalisation | Discharge | Criteria | Onset | |
| XX-XXX | XX | Male/Female | XXXX | DD-MMM-YYYY | DD-MMM-YYYY | Yes/No | DD-MMM-YYYY | DD-MMM-YYYY | XXXX | DD-MMM-YYYY | xxxx |
| XX-XXX | XX | Male/Female | XXXX | DD-MMM-YYYY | DD-MMM-YYYY | Yes/No | DD-MMM-YYYY | DD-MMM-YYYY | XXXX | DD-MMM-YYYY | XXXX |
| XX-XXX | XX | Male/Female | XXXX | DD-MMM-YYYY | DD-MMM-YYYY | Yes/No | DD-MMM-YYYY | DD-MMM-YYYY | XXXX | DD-MMM-YYYY | XXXX |
| XX-XXX | XX | Male/Female | XXXX | DD-MMM-YYYY | DD-MMM-YYYY | Yes/No | DD-MMM-YYYY | DD-MMM-YYYY | XXXX | DD-MMM-YYYY | XXXX |
| XX-XXX | XX | Male/Female | XXXX | DD-MMM-YYYY | DD-MMM-YYYY | Yes/No | DD-MMM-YYYY | DD-MMM-YYYY | XXXX | DD-MMM-YYYY | xxxx |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

## Listing 16.3.3.1 Listing of Patients Haematology (WHOLE BLOOD)

| Patient | | Blood Sample | If No, Specify | Date and Time of blood | | | | | If Abnormal CS, describe |
|---|---|---|---|---|---|---|---|---|---|
| Number | Visit | Collected | Reason | Sample | <b>Parameters</b> | Result | Unit | Normal/Abnormal NCS | the abnormality# |
| xx-xxx | XXXX | Yes/No | xxxx | DD-MMM-YYYY/HH:MM | xxxx | XXXX | XXXX | Normal/Abnormal NCS | xxxx |
| xx-xxx | XXXX | Yes/No | xxxx | DD-MMM-YYYY/HH:MM | XXXX | XXXX | XXXX | Normal/Abnormal NCS | xxxx |
| XX-XXX | XXXX | Yes/No | xxxx | DD-MMM-YYYY/HH:MM | xxxx | XXXX | XXXX | Normal/Abnormal NCS | xxxx |
| XX-XXX | XXXX | Yes/No | xxxx | DD-MMM-YYYY/HH:MM | XXXX | XXXX | XXXX | Normal/Abnormal NCS | xxxx |
| XX-XXX | XXXX | Yes/No | XXXX | DD-MMM-YYYY/HH:MM | XXXX | XXXX | XXXX | Normal/Abnormal NCS | xxxx |



| Document Title: | Document ID: | BP04-01 |
|------------------------------|-----------------|-------------|
| Statistical Affailysis Plaff | Effective Date: | 25-Nov-2021 |

## Listing 16.3.3.2. Listing of Patients Clinical chemistry (Plasma / Serum)

| Patient | | Blood Sample | If No, Specify | Date and Time of blood | | | | | If Abnormal CS, describe |
|---|---|---|---|---|---|---|---|---|---|
| Number | Visit | Collected | Reason | Sample | Parameters | Result | Unit | Normal/Abnormal NCS | the abnormality# |
| xx-xxx | XXXX | Yes/No | xxxx | DD-MMM-YYYY/HH:MM | xxxx | XXXX | XXXX | Normal/Abnormal NCS | xxxx |
| XX-XXX | XXXX | Yes/No | XXXX | DD-MMM-YYYY/HH:MM | xxxx | XXXX | XXXX | Normal/Abnormal NCS | xxxx |
| XX-XXX | XXXX | Yes/No | XXXX | DD-MMM-YYYY/HH:MM | XXXX | XXXX | XXXX | Normal/Abnormal NCS | xxxx |
| XX-XXX | XXXX | Yes/No | XXXX | DD-MMM-YYYY/HH:MM | XXXX | XXXX | XXXX | Normal/Abnormal NCS | xxxx |
| XX-XXX | XXXX | Yes/No | XXXX | DD-MMM-YYYY/HH:MM | XXXX | XXXX | XXXX | Normal/Abnormal NCS | xxxx |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

## Listing 16.3.3.3. Listing of Patients Urinalysis (Dipstick)

| Patient | | Urine Sample | If No, Specify | Date and Time of Urine | | | | | If Abnormal CS, describe the |
|---|---|---|---|---|---|---|---|---|---|
| Number | Visit | Collected | Reason | Sample | Parameters | Result | Unit | Normal/Abnormal NCS | abnormality# |
| XX-XXX | XXXX | Yes/No | xxxx | DD-MMM-YYYY/HH:MM | XXXX | XXXX | XXXX | Normal/Abnormal NCS | xxxx |
| XX-XXX | XXXX | Yes/No | XXXX | DD-MMM-YYYY/HH:MM | XXXX | XXXX | XXXX | Normal/Abnormal NCS | xxxx |



| Document Title: | Document ID: | BP04-01 |
|------------------------------|-----------------|-------------|
| Statistical Affailysis Plaff | Effective Date: | 25-Nov-2021 |

## Listing 16.3.4. Listing of Patients Electrocardiogram (ECG)

| Patient | | ECG | If No, Specify | | | | | | If Abnormal CS, describe the |
|---|---|---|---|---|---|---|---|---|---|
| Number | Visit | Performed | Reason | Date and Time of ECG | Parameter | Result | Unit | Normal/Abnormal NCS | abnormality# |
| xx-xxx | XXXX | Yes/No | xxxx | DD-MMM-YYYY/HH:MM | xxxx | XXXX | XXXX | Normal/Abnormal NCS | xxxx |
| XX-XXX | XXXX | Yes/No | XXXX | DD-MMM-YYYY/HH:MM | xxxx | XXXX | XXXX | Normal/Abnormal NCS | xxxx |
| XX-XXX | XXXX | Yes/No | XXXX | DD-MMM-YYYY/HH:MM | xxxx | XXXX | XXXX | Normal/Abnormal NCS | xxxx |
| XX-XXX | XXXX | Yes/No | XXXX | DD-MMM-YYYY/HH:MM | XXXX | XXXX | XXXX | Normal/Abnormal NCS | xxxx |
| XX-XXX | XXXX | Yes/No | XXXX | DD-MMM-YYYY/HH:MM | XXXX | XXXX | XXXX | Normal/Abnormal NCS | xxxx |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## Listing 16.3.5. Listing of Patients Vital Signs

| Patient | | Vital Signs | If No, Specify | Date of Vital | | | | If Abnormal CS, describe the |
|---|---|---|---|---|---|---|---|---|
| Number | Visit | Collected | Reason | Signs | Parameter | Result | Normal/Abnormal NCS | abnormality# |
| xx-xxx | XXXX | Yes/No | xxxx | DD-MMM-YYYY | xxxx | XXXX | Normal/Abnormal NCS | xxxx |
| XX-XXX | XXXX | Yes/No | XXXX | DD-MMM-YYYY | xxxx | XXXX | Normal/Abnormal NCS | xxxx |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## Listing 16.3.6. Listing of Patients Physical Examination

| Patient | | Physical Examination | If No, Specify | Date of Physical | Seq. | | | If Abnormal CS, describe |
|---|---|---|---|---|---|---|---|---|
| Number | Visit | Performed | Reason | Examination | No. | System | Normal/Abnormal NCS | the abnormality# |
| XX-XXX | XXXX | Yes/No | xxxx | DD-MMM-YYYY | XX | XXXX | Normal/Abnormal NCS | xxxx |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## Listing 16.3.7. Listing of Patients Other Assessment

| Patient | | Hypoglycemic | Urinary Tract | Gental Tract | Volume | Diabetic | Renal | Hospitalization |
|---|---|---|---|---|---|---|---|---|
| Number | Visit | Events | Infection | Infection | depletion | Ketoacidosis | Events | for Heart Failure |
| XX-XXX | XXXX | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## Listing 16.3.8.1. Listing of Patients Urinary Tract Infection

| Patient | | Urine Sample | Date and Time of Sample | Patient confirmed with | | Urinary Tract | | | |
|---|---|---|---|---|---|---|---|---|---|
| Number | Visit | obatianed for culture | Collection | Urinnary tract Infection | Cystitis | Infection | Pyelonephritis | Prostatitis | Other |
| xx-xxx | XXXX | Yes/No | DD-MMM-YYYY/HH:MM | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| XX-XXX | XXXX | Yes/No | DD-MMM-YYYY/HH:MM | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## Listing 16.3.8.2. Listing of Patients Genital Tract Infection

| Patient | | Urine Sample obatianed | If No, specify | Date and Time of Sample | Patient confirmed with | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Number | Visit | for genital swab | reason | Collection | Gential tract Infection | Vaginitis | Vulvoviginitis | Vulvitis | Balantis |
| xx-xxx | XXXX | Yes/No | xxxx | DD-MMM-YYYY/HH:MM | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |
| XX-XXX | XXXX | Yes/No | XXXX | DD-MMM-YYYY/HH:MM | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Listing 16.3.8.3. Listing of Patients Volume Depletion

| Patient Number | Visit | Patient at high risk of Volume Depletion | Dehydrtion | Hypovolemia | Hypptensio |
|---|---|---|---|---|---|
| XX-XXX | XXXX | Yes/No | Yes/No | Yes/No | Yes/No |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Listing 16.3.8.4. Listing of Patients Diabetic Ketoacidosis

| | | Patient conformed | Date of DKA | Medication Taken | Action Taken with Investigation |
|---|---|---|---|---|---|
| Patient Number | Visit | with DKA | Conformation | for the Events | Product |
| XX-XXX | XXXX | Yes/No | DD-MMM-YYYY | Yes/No | Discontinued/ Temporary Stopped |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## Listing 16.3.8.5. Listing of Patients Renal Events

| | | Renal Event | Doubling of serum | | |
|---|---|---|---|---|---|
| Patient Number | Visit | Occurred | creatinine | Dialysis | Renal transpiantion |
| XX-XXX | XXXX | Yes/No | Yes/No | Yes/No | Yes/No |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Listing 16.3.8.6. Listing of Patients Hospitalization for Heart Failure

| | | Patient admitted to the hospital with | Patient hospitalized for nore |
|---|---|---|---|
| Patient Number | Visit | Primary diagnosis of Heart Failure | than 24 hours |
| XX-XXX | XXXX | Yes/No | Yes/No |
| XX-XXX | XXXX | Yes/No | Yes/No |
| XX-XXX | XXXX | Yes/No | Yes/No |
| XX-XXX | XXXX | Yes/No | Yes/No |
| XX-XXX | XXXX | Yes/No | Yes/No |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Listing 16.3.9.1. Listing of Patients Concomitant Medications

| | | Patient Take any other concomitant | Patient Take any other concomitant |
|---|---|---|---|
| Patient Number | Visit | medication during Visit | medication since last visit |
| XX-XXX | XXXX | Yes/No | Yes/No |
| XX-XXX | XXXX | Yes/No | Yes/No |
| XX-XXX | XXXX | Yes/No | Yes/No |
| XX-XXX | XXXX | Yes/No | Yes/No |
| XX-XXX | XXXX | Yes/No | Yes/No |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## Listing 16.3.9.2. Listing of Patients Concomitant Medication

| Patient | Patient Receive Any | Seq. | Medication | Start Date / | | | Dose | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Number | Concomitant Medication | No | name | Stop date | Ongoing | Indication | Form | Dose | unit | Route | Frequency |
| | | | | DD-MMM-YYYY/ | | | | | | | _ |
| XX-XXX | Yes/No | XX | XXX | DD-MMM-YYYY | XXXX | xxxx | XXXX | XXXX | XXXX | XXXX | xxxx |
| | | | | DD-MMM-YYYY/ | | | | | | | |
| XX-XXX | Yes/No | XX | XXX | DD-MMM-YYYY | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | xxxx |
| | | | | DD-MMM-YYYY/ | | | | | | | |
| XX-XXX | Yes/No | XX | XXX | DD-MMM-YYYY | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX |
| | | | | DD-MMM-YYYY/ | | | | | | | |
| XX-XXX | Yes/No | XX | XXX | DD-MMM-YYYY | XXXX | xxxx | XXXX | XXXX | XXXX | XXXX | xxxx |
| | | | | DD-MMM-YYYY/ | | | | | | | |
| XX-XXX | Yes/No | XX | XXX | DD-MMM-YYYY | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX |